CLINICAL TRIAL: NCT06596785
Title: Investigation and Early Risk Prediction of Acute Kidney Injury Caused by Iodinated Contrast Agents: Development of CI-AKIDPi Model Based on Interpretable Deep Learning
Brief Title: Risk Factors and Deep Learning Model for CI-AKI
Status: Active, not recruiting | Type: Observational
Sponsor: Xiao Li，MD (Other)
Responsible Party: Sponsor-Investigator, Xiao Li，MD, Associate professor of pharmacy, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: LCYX-LX-20240101
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contrast-associated acute kidney injury (CI-AKI) is a sudden and significant decline in renal function resulting from the use of a contrast agent.

DETAILED DESCRIPTION:
Contrast-associated acute kidney injury (CI-AKI) is a sudden and significant decline in renal function resulting from the use of a contrast agent. Despite the frequent use of iodinated contrast agents in medical investigations, predictive models for CI-AKI are scarce. This study aimed to construct and validate interpretable deep learning models for the early risk prediction of acute kidney injury (AKI) associated with iodinated contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* patients who received iodinated contrast agents during hospitalization
* age ≥ 18 years
* hospitalization length ≥ 48 hours
* at least two serum creatinine tests during hospitalization

Exclusion Criteria:

* patients with stage 4 or 5 chronic kidney disease prior to admission
* patients undergoing hemodialysis, hemofiltration or peritoneal before admission
* a history of nephrectomy or kidney transplantation during hospitalization
* incomplete clinical information
* Serum creatinine always ≤ 40 μmol/L during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
AKI | Completed through study, up to half a year
  During the patient's hospitalization, acute kidney injury occurred after the use of Iodinated contrast media

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Lii, Principal Investigator — Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China